CLINICAL TRIAL: NCT01083082
Title: Physical Exercise, Fitness and Dietary Pattern and Theirs Relationship With Blood Pressure Circadian Pattern, Augmentation Index and Endothelial Dysfunction Biological Markers. (EVIDENT Study)
Brief Title: Lifestyles and Endothelial Dysfunction
Acronym: EVIDENT
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: PS09/00233
Record Dates: First submitted 2010-03-06; First posted 2010-03-09 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: lifestyles; diet; exercise; central blood pressure; arterial stiffness; endothelial dysfunction; Healthy people
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Objectives: To analyze the relationship of physical activity, fitness, energy intake and dietary pattern with the circadian pattern of blood pressure, central and peripheral blood pressure pulse wave velocity and biological markers of endothelial dysfunction in active and sedentary people without atherosclerotic disease.

DETAILED DESCRIPTION:
Objectives: To analyze the relationship of physical activity, fitness, energy intake and dietary pattern with the circadian pattern od blood pressure, central and peripheral blood pressure pulse wave velocity and biological markers of endothelial dysfunction in active and sedentary people without atherosclerotic disease.

Methods:

Design: Cross- sectional study 1ª step of clinical trial later. Project multicentric with seis research groups.

Subjects: From subjects of PEPAF project cohort, that remain in last control 3105 (1.163 active and sedentary 1942) and 2346 were excluded for actives. By Random sampling included 352 subjects who remained sedentary, 588 who have become active and 560 of which were excluded for being active in baseline assessment, a total of 1,200. Each of the six groups included 250 subjects.

Measurements: We evaluated height, weight, abdominal perimeter, blood pressure clinic, ambulatory blood pressure with Radial pulse wave acquisition device (BPro), central blood pressure, (aortic) and Augmentation index with Pulse Wave Application Software (A-Pulse) and Sphigmo cor System Px (Pulse Wave Analysis), pulse wave velocity (PWV) with Sphigmo cor System Px (Pulse Wave velocity), nutritional pattern with a food consumption survey, physical activity 7 Par-day questionnaire and the accelerometer (MTI/CSA 7164) and physical fitness with cicloergometro (PWC170) and endothelial dysfunction biomarkers (endoglin and osteoprotegerin).

ELIGIBILITY:
Inclusion Criteria:

* Healthy people
* Ages 20-80 years old

Exclusion Criteria:

* Cardiovascular disease
* Respiratory failure
* Patient ends
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people 20-80 aged that visit their family doctor and accept be involved in study from six Spanish cities
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2010-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Physical activity | December, 1 2014

SECONDARY OUTCOMES:
diet | december, 1 2014

OTHER OUTCOMES:
blood pressure | december 1, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Luis Garcia, MD, Principal Investigator — Fundacion para la investigación y formacion en ciencias de la salud
Locations (1):
- Luis Garcia Ortiz, Salamanca, Spain

REFERENCES:
- [Derived] Garcia-Hermoso A, Martinez-Vizcaino V, Recio-Rodriguez JI, Diez-Fernandez A, Gomez-Marcos MA, Garcia-Ortiz L; Evident Group. Abdominal obesity as a mediator of the influence of physical activity on insulin resistance in Spanish adults. Prev Med. 2016 Jan;82:59-64. doi: 10.1016/j.ypmed.2015.11.012. Epub 2015 Nov 19. PMID 26601643
- [Derived] Garcia-Hermoso A, Martinez-Vizcaino V, Sanchez-Lopez M, Recio-Rodriguez JI, Gomez-Marcos MA, Garcia-Ortiz L; EVIDENT Group. Moderate-to-vigorous physical activity as a mediator between sedentary behavior and cardiometabolic risk in Spanish healthy adults: a mediation analysis. Int J Behav Nutr Phys Act. 2015 Jun 20;12:78. doi: 10.1186/s12966-015-0244-y. PMID 26437664
- [Derived] Patino-Alonso MC, Recio-Rodriguez JI, Magdalena-Belio JF, Gine-Garriga M, Martinez-Vizcaino V, Fernandez-Alonso C, Arietaleanizbeaskoa MS, Galindo-Villardon MP, Gomez-Marcos MA, Garcia-Ortiz L; EVIDENT Group. Clustering of lifestyle characteristics and their association with cardio-metabolic health: the Lifestyles and Endothelial Dysfunction (EVIDENT) study. Br J Nutr. 2015 Sep 28;114(6):943-51. doi: 10.1017/S0007114515002500. Epub 2015 Aug 13. PMID 26268844
- [Derived] Garcia-Hermoso A, Martinez-Vizcaino V, Recio-Rodriguez JI, Sanchez-Lopez M, Gomez-Marcos MA, Garcia-Ortiz L; EVIDENT Group. Sedentary behaviour patterns and carotid intima-media thickness in Spanish healthy adult population. Atherosclerosis. 2015 Apr;239(2):571-6. doi: 10.1016/j.atherosclerosis.2015.02.028. Epub 2015 Feb 23. PMID 25733329
- [Derived] Gomez-Marcos MA, Recio-Rodriguez JI, Patino-Alonso MC, Agudo-Conde C, Lasaosa-Medina L, Rodriguez-Sanchez E, Maderuelo-Fernandez JA, Garcia-Ortiz L; EVIDENT Group. Relationship between objectively measured physical activity and vascular structure and function in adults. Atherosclerosis. 2014 Jun;234(2):366-72. doi: 10.1016/j.atherosclerosis.2014.02.028. Epub 2014 Mar 18. PMID 24742874
- [Derived] Garcia-Ortiz L, Recio-Rodriguez JI, Schmidt-Trucksass A, Puigdomenech-Puig E, Martinez-Vizcaino V, Fernandez-Alonso C, Rubio-Galan J, Agudo-Conde C, Patino-Alonso MC, Rodriguez-Sanchez E, Gomez-Marcos MA; EVIDENT Group. Relationship between objectively measured physical activity and cardiovascular aging in the general population--the EVIDENT trial. Atherosclerosis. 2014 Apr;233(2):434-440. doi: 10.1016/j.atherosclerosis.2014.01.021. Epub 2014 Jan 24. PMID 24530775
- [Derived] Garcia-Ortiz L, Recio-Rodriguez JI, Puig-Ribera A, Lema-Bartolome J, Ibanez-Jalon E, Gonzalez-Viejo N, Guenaga-Saenz N, Agudo-Conde C, Patino-Alonso MC, Gomez-Marcos MA; EVIDENT Group. Blood pressure circadian pattern and physical exercise assessment by accelerometer and 7-day physical activity recall scale. Am J Hypertens. 2014 May;27(5):665-73. doi: 10.1093/ajh/hpt159. Epub 2013 Aug 24. PMID 23975330
- [Derived] Garcia-Ortiz L, Recio-Rodriguez JI, Martin-Cantera C, Cabrejas-Sanchez A, Gomez-Arranz A, Gonzalez-Viejo N, Iturregui-San Nicolas E, Patino-Alonso MC, Gomez-Marcos MA; EVIDENT Group. Physical exercise, fitness and dietary pattern and their relationship with circadian blood pressure pattern, augmentation index and endothelial dysfunction biological markers: EVIDENT study protocol. BMC Public Health. 2010 May 6;10:233. doi: 10.1186/1471-2458-10-233. PMID 20459634